CLINICAL TRIAL: NCT04031287
Title: A Prospective Natural History Study of Patients With Rhizomelic Chondrodysplasia Punctata (RCDP)
Brief Title: RCDP Natural History Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: MED-LIFE DISCOVERIES LP (Industry)
Responsible Party: Sponsor
Other Study IDs: MLD_CT1.0
Record Dates: First submitted 2019-06-13; First posted 2019-07-24 (Actual); Last update posted 2019-08-02 (Actual); Status verified 2019-08

CONDITIONS: Rhizomelic Chondrodysplasia Punctata
MeSH Terms: conditions — Chondrodysplasia Punctata, Rhizomelic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 18 Months
Biospecimen Retention: Samples With DNA — Blood samples
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A prospective, longitudinal observational trial in patients with RCDP. Study participants will be evaluated at baseline and approximately every 6 months by the study team. Quality of life, physiologic and functional measurements will be performed. In addition, audiologic recordings and other surveys will be completed at home by parents beginning at baseline and every 3-6 months thereafter.

DETAILED DESCRIPTION:
Rhizomelic chondrodysplasia punctata (RCDP) is a group of rare diseases that have no known cure. It is a genetic disorder characterized by mutations in the Peroxisomal Biogenesis Factor 7 (PEX7) gene (RCDP1), Glyceronephosphate O-acyltransferase (GNPAT) gene (RCDP 2), Alkylglycerone phosphate synthase (AGPS) gene (RCDP3), Fatty Acyl-CoA Reductase 1 (FAR1) gene (RCDP4) or Peroxisomal Biogenesis Factor 7 (PEX7) gene (RCDP5) all coding for peroxisomal proteins which result in defective synthesis of plasmalogens. Hence, severely decreased levels of ethanolamine plasmalogens (PlsEtn), the most common tissue plasmalogen, is both the biochemical hallmark and the primary cause of pathology for all RCDP groups. To treat RCDP, a plasmalogen replacement is under development. Before this therapeutic or any therapeutic for RCDP can be tested for efficacy in the clinic, a thorough understanding of the natural progression of the disease is required. Without this information it would be impossible to determine whether the drug was effectively improving the disease course. Classical, or severe, is the most common form of RCDP and presents in the neonatal period. It is clinically characterized by a skeletal dysplasia as seen by symmetrical rhizomelic shortening of the long bones. Chondrodysplasia is also present with premature calcification of epiphyseal cartilage (punctata), delayed calcification of vertebral bodies and mineralization of cartilaginous structures which do not normally ossify, such as the larynx, trachea and intervertebral discs. Additionally patients display dysmorphic facial features, bilateral cataracts, cognitive deficits and severe growth and psychomotor delays. Shortened life expectancy is common to RCDP patients; however survival varies widely. For the classical form, of those individuals who survive the first month of life, 50% will survive until 6 years of age with nearly all succumbing to the disease by adolescence. The majority of deaths are secondary to respiratory problems5. The chronic respiratory compromise is due to the skeletal defects, as well as the direct effect of plasmalogen deficiency on lung cellular function. Patients with less severe phenotypes can lack rhizomelia, and have less severe growth and developmental delays. The disease phenotype varies considerably and correlates directly with PlsEtn abundance.

STUDY RATIONALE Determining the appropriate measurable endpoints are as important as having a viable therapeutic strategy for a clinical trial. In a disease like RCDP, endpoints must be sensitive enough to measure subtle changes in the course of the disease and also be meaningful to the process of pathogenesis. Assessment of a RCDP treatment trial is a complex task as RCDP clinical trajectory might be influenced by the disease severity, age and care that the patient receives etc. Moreover, although measurement scales exist for such diseases as Cerebral Palsy to assess the severity of the disease, RCDP does not have such universally accepted overall set of measures that assess patient's developmental, functional, psychosocial, neurological, skeletal, and respiratory functions as a whole. Lack of such grading scales is a hindrance to evaluate the progress of a clinical trial in a complex and severe disease as RCDP. In a disease like RCDP, more than a complete cure, a functional improvement in patient's life could be considered as efficacious.

The other issue in a rare disease clinical trial design is the comparator to which the effect of treatment can be compared. Ethical considerations preclude having a placebo control and a more appropriate comparator is a non-concurrent control group. Therefore, longitudinal assessments are required to determine the inherent variability in functional measures and characterize the disease trajectory. To this end, we have designed an on-going longitudinal observational trial with assessments every 3-6 months to characterize RCDP and its disease course.

Overarching goal is to determine the longitudinal and natural trajectory of disease state in patients with RCDP by assess the quality of life, physiologic and functional measures.

Specific measurements will include:

* Medical and surgical history
* Anthropometric measurements
* Vital signs
* Physical examination
* Observational pain assessment
* Musculoskeletal system assessment
* Nerve conduction studies
* Non-invasive pulmonary function tests

  * Impulse Oscillometry System
  * Pneumotachography
  * Respiratory Inductance Plethysmography
* 4 hour EEG
* DEXA
* Questionnaire assessment of:

  * Iowa Fatigue Scale
  * Pediatric Pain Scale
  * NCCPC-R (Pain Scale)
  * Infant Gastrointestinal Symptom Questionnaire
  * Pediatric Assessment Scale for Severe Feeding Problems
* LENA
* Parental written logs (over 2 days)

  * Activity
  * Pain
  * Seizure
* Blood Assessments

  * Plasmalogen and Lipids
  * Complete Blood Count
  * Comprehensive Metabolic Panel
  * Genetic Testing (if not available from history)

STUDY DESIGN

As described above, clinical characteristics of RCDP encompass a wide range of signs, symptoms, physiological, functional and structural abnormalities all of which must be taken in to account when assessing a patient's progress. The major systems affected are the skeletal system (severe and symmetrical shortening of proximal long bones, stippled epiphyses, dysmorphia and contractures), neurophysiological (seizures), neuromuscular and psychomotor abnormalities, respiratory, growth and developmental and daily function. Many of these symptoms can be characterized by standard tests that are in clinical or research use. Other assessments, such as the quality of life, require the development of novel tools which will be implemented once they have been validated. Assessing each domain in its own right will provide the best indication of efficacy on an individual basis.

Domain specific milestones as described here will increase the sensitivity in assessing treatment specific effects. Acute clinically evident improvements brought about by plasmalogen replacement therapy are expected to be subtle. The earliest improvements are anticipated to be improvements in membrane-related functions such as improved neurotransmission, improved neuromuscular function, improved GI function, increase growth rates and better lung health. Functionally, we anticipate that primary and immediate improvements will be evident in motor function, frequency of seizures, frequency of pulmonary infections and improved quality of life. Improvements in other systems and function are anticipated to arise later in a gradual manner. Consequently, assessment of each of these domains as well as an assessment of quality of life and measures of functionality are needed to estimate therapeutic benefits accurately.

The study is intended to be on-going, allowing for longitudinal assessment of RCDP. In- hospital assessments will be completed approximately every 6 months, based on availability of scheduling and patients' health. In home audiologic recordings will take place after each study visit along with parent completed logs. In home surveys will be distributed every 3 months to the caregiver.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of RCDP age range 6 months to 21 years
* A clinical diagnosis of RCDP confirmed with biochemical parameters defined as C16:0 plasmalogen level of less than or equal to 0.75 of the lower limit of the normal reference range AND normal very long chain fatty acid levels.

Exclusion Criteria:

* Disease severity: The study physician will decide whether the child is too ill to travel due to chronic or acute severe cardiac or respiratory compromise.
* Guardian or a care-giver who is not available or not capable of providing accurate information about the patient.
* Involvement in any other clinical trial.

Ages: 6 Months to 21 Years | Sex: All
Age Groups: Child, Adult
Study Population: Patients with a diagnosis of RCDP are eligible.
Sampling Method: Non-Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2019-06-18 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
Medical History | 18 months
  History collection will be obtained from parents/caretakers and medical records which will be provided or subsequently obtained in a HIPAA compliant manner.
Body Temperature | 18 months
  Temperature will be recorded using standard clinical methodology and reported in degrees Celsius.
Respiratory Rate | 18 months
  Respiratory rate will be determined by counting number of breaths per minute
Heart Rate | 18 months
  Heart rate will be reported as beats per minute
Blood pressure | 18 months
  Systolic and diastolic pressure will be reported in mmHG
Physical Examination: General Appearance | 18 months
  Reported as "Normal, Abnormal or Not Done". If abnormal, comments will be provided.
Physical Examination: Head, Eyes, Ears, Nose and Throat | 18 months
  Reported as "Normal, Abnormal or Not Done". If abnormal, comments will be provided.
Physical Examination: Cardiovascular | 18 months
  Reported as "Normal, Abnormal or Not Done". If abnormal, comments will be provided.
Physical Examination: Dermatologic | 18 months
  Reported as "Normal, Abnormal or Not Done". If abnormal, comments will be provided.
Physical Examination: Lymphatic | 18 months
  Reported as "Normal, Abnormal or Not Done". If abnormal, comments will be provided.
Physical Examination: Respiratory | 18 months
  Reported as "Normal, Abnormal or Not Done". If abnormal, comments will be provided.
Physical Examination: Gastrointestinal | 18 months
  Reported as "Normal, Abnormal or Not Done". If abnormal, comments will be provided.
Physical Examination: Genitourinary | 18 months
  Reported as "Normal, Abnormal or Not Done". If abnormal, comments will be provided.
Physical Examination: Neurologic System | 18 months
  Reported as "Normal, Abnormal or Not Done". If abnormal, comments will be provided.
Physical Examination: FLACC Behavioural Scale | 18 months
  The standardized FLACC (Faces, Legs, Activity, Consolability) questionnaire will be performed and the score reported.
Anthropometric Measurement: Length/Height | 18 months
  Height (Length) will be reported in centimetres
Anthropometric Measurement: Weight | 18 months
  Weight will be reported in kg
Anthropometric Measurement: Head Circumference | 18 months
  Head Circumference will be reported in cm
Anthropometric Measurement: Chest Circumference | 18 months
  Chest Circumference will be reported in cm
Anthropometric Measurement: Abdominal Circumference | 18 months
  Abdominal Circumference will be reported in cm
Observational pain assessment | 18 months
  Frequency and severity of patient exhibited pain symptoms will be evaluated with two parent-completed questionnaires, The Non-Communicating Children's Pain Checklist- Revised (NCCPC-R) and the Pediatric Pain Scale (PPS)19 (Appendix G). The NCCPC-R is a 7 domain questionnaire that is validated for assessment of pain in children aged 3-18 years who have cognitive and communication impairments. The PPS has 20 domains with a rating scale for each which is also designed to assess symptoms of pain in individuals with communication impairment. Both questionnaires will be completed during the study visits 2 hours after the end of the first morning feed. In addition, the NCCPC-R will be completed by the family 3 months after each visit at the same time interval after the first morning feed.
Musculoskeletal system assessment | 18 months
  Musculoskeletal evaluations will be done together by a physiatrist and physical therapy. These assessments will include: assessments of strength, endurance, functional movement and control of extremities, head/neck and trunk. Assessment of muscle tone and passive and active joint range of motion will be made both qualitative and quantitatively for each major joint. Assessment of cognitive engagement will also be made. To assess the motor function and its changes over time, we propose to use Gross Motor Function Measures (GMFM-88), which is a freely available tool validated to evaluate motor skills in cerebral palsy and Down syndrome.
Nerve conduction | 18 months
  Patients will be placed in a supine position and electrodes will be placed over the hypothenar eminence, 5th digit and dorsal hand. Stimulations will be done at the wrist and above and below the elbow. These electrodes will be connected to the Natus UltraPro S100 machine. This unit will measure nerve conduction for motor and sensory components. The evaluation will assess nerve latencies, compound motor unit and sensory nerve action potential amplitudes and nerve conduction velocities. These values will be compared to age adjusted normal values for the ulnar nerve.
Pulmonary function | 18 months
  A combination of Impulse oscillometry system (IOS), Pneumotachography (PNT) and Respiratory Inductance Plethysmography (RIP) will be used to derive pulmonary indices comparable to spirometry.
Seizure status by EEG | 18 months
  Assessments of brain electrical and seizure activity will take place through electroencephalograms (EEGs) at each study visit. Each EEG will last 4 hours and will be scheduled to optimally include both awake and sleep phases. Using the 10-20 International System, the patient's head will be measured and marked for proper electrode placement. Heart rate and rhythm are monitored throughout the EEG by placement of two electrocardiogram electrodes. Electrical activity is then recorded along with a video feed using the Nicolet NicOne acquisition and Xltek brain monitor machines.
Bone Density and Body Composition by DEXA | 18 months
  The DEXA scans will be performed in the Medical Imaging Department of Nemours/A.I. duPont Hospital for Children on a Hologic Discovery A QDR bone densitometer (Hologic, Inc., Bedford, MA). Subjects will remove all clothing with metal components prior to DEXA scan to eliminate any possible imaging artifacts; a hospital gown will be provided to the subjects. Standard positioning techniques will be used to acquire the scans. Body sites measured will include the whole body, lumbar spine, and lateral distal femurs of both legs. The following variables will be collected from each scan: bone mineral density (BMD), bone mineral content (BMC), and bone area.
Plasmalogen Level | 18 months
  A 100 ul aliquot of the separated serum will be stored at -80 °C and subsequently shipped to Med-Life Discoveries by priority overnight shipment in dry ice. Analyses will include levels of phosphoethanolamines, vinylacylglycerol (VAG), alkylacylglycerol (AAG) and results reported as quantitative concentrations for each metabolite.
Clinical Chemistry | 18 months
  Serum will be processed locally for complete blood count (CBC) and standard comprehensive metabolic profile with phosphorus (CMP with PO4).
Fatigue status | 18 months
Gastrointestinal and Feeding status | 18 months
  To assess level of dysfunction in swallowing, a parent report measure, the Pediatric Assessment Scale for Severe Feeding Problems, designed to assess progress in the development of oral eating skills for children who need prolonged tube feeding will be used. The total score will be used as a quantifiable measure. This questionnaire will be completed during each study visit as well as at home 3 months after each visit. This 13 question interview provides a total score which indicates the level of GI symptom burden.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Bober, MD, Principal Investigator — The Nemours Foundation
Locations (1):
- Alfred I. DuPont Hospital for Children, Wilmington, Delaware, United States